CLINICAL TRIAL: NCT04602195
Title: Responsiveness and Validation Study of MFM-32 in SMA Patients Treated With Nusinersen: NusiMFM
Brief Title: Responsiveness and Validation Study of MFM-32 in SMA Patients Treated With Nusinersen
Acronym: NusiMFM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0875
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-04

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy, Motor Function Measure,Nusinersen
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Motor Function Measure (MFM), a reliable tool assessing motor function and its progression in most neuromuscular diseases, is widely used in France in many teams. It can be used regardless of the severity of the motor impairment or the ambulatory status of the patient, allowing its use throughout the whole follow-up period of the patient, even in case of the loss of walking. Two versions of the MFM exist, one composed of 32 items originally validated for patients from 6 years old (MFM-32) and a shorter version composed of 20 items originally validated for patients between 2 and 6 years old (MFM-20).

In order to prove the possible use of MFM-32 as early as the age of 2 years to validly and reliably monitor the evolution of the motor function of children treated with Nusinersen, we propose in this project to study the sensitivity to treatment-induced change of MFM-32 and the validity of the scale in this population.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls with Type 1 or 2 Spinal Muscular Atrophy, genetically confirmed
* Aged 2 to 6 years old
* Treated by Nusinersen for at least two months
* With parental assent

Exclusion Criteria:

* Patients with associated cognitive impairment making impossible evaluation of motor function
* Patients participating to a clinical study with a potential effect on their motor function.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * Boys and girls with Type 1 or 2 Spinal Muscular Atrophy, genetically confirmed
  * Aged 2 to 6 years old
  * Treated by Nusinersen for at least two months
  * With parental assent
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
MFM-32 responsiveness | 1 Year after the first MFM-32 assessment
  Responsiveness of MFM-32 in comparison to PGIC. The responsiveness sensitivity to change indexes considered will be the effect size (ES) amplitude and the Standardized Response Mean (SRM)

CONTACTS AND LOCATIONS:
Overall Officials: Laure Le Goff, MD, Principal Investigator — L'Escale, Service central de rééducation pédiatrique
Locations (10):
- France (10):
  - Service de neuropédiatrie et neurochirurgie de l'enfant Centre de Référence des Maladies Neuromusculaires AOC CHU d'Angers, Angers
  - Centre de Référence des maladies neuromusculaires Centre Hospitalier Régional Universitaire de Brest, Brest
  - L'Escale, Service central de rééducation pédiatrique Hospices Civils de Lyon Hôpital Mere Enfant, Bron
  - Service de génétique médicale Pôle de Pédiatrie CHU Estaing, Clermont-Ferrand
  - Service de Neurologie et réanimation pédiatriques, Garches
  - Apf Esean, Nantes
  - Institut I-Motion - Centre de recherche pédiatrique en pathologies neuromusculaires, Paris
  - Service de pédiatrie CHU de Saint-Etienne, Saint-Priest-en-Jarez
  - Service de Neuropédiatrie CHU de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - Unité de Neurologie Pédiatrique Centre de Référence Maladies NeuroMusculaires Hôpital des Enfants CHU Toulouse, Toulouse